CLINICAL TRIAL: NCT05103839
Title: A Pilot Study Yoga for Caregivers and Persons With Dementia
Brief Title: Yoga for Caregivers and Persons With Dementia
Acronym: YCPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00077146
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-12

CONDITIONS: Dementia
Keywords: dyad; caregiver; yoga; dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga for Caregivers and Persons With Dementia (Experimental): Persons With Dementia and their caregivers will participate in up to 20 group yoga classes.
  Interventions: Behavioral: Gentle Yoga

INTERVENTIONS:
Behavioral: Gentle Yoga — Yoga classes are twice a week for up to 10 weeks with a trained yoga instructor at a location in the community. Classes will last up to 75 minutes.

SUMMARY:
The purpose of this research is to determine the feasibility and acceptability of yoga classes for persons living with dementia (PLWD) and their care partners. A secondary aim of this study is to examine the impact of yoga on caregiver burden.

DETAILED DESCRIPTION:
Participants will be recruited from the D-Care Study in dyads. Both the caregiver and person with dementia must agree to participate. Screening will be done either in clinics or by telephone in the participants' homes. The intervention will be conducted in community facilities and participants' homes. The sample size will consist of 10 caregiver/person with dementia dyads. This number was chosen to provide evidence of feasibility of conducting yoga classes with dyads.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers: Providing unpaid care to a family member of friend diagnosed Alzheimer's Disease and Alzheimer's Disease Related Dementias (ADRD)
* Persons with dementia: A diagnosis of dementia; live in the community (assisted living facility is allowed); cognitively able to participate in yoga as determined by study staff

Exclusion Criteria:

* Non-English-speaking; and practicing yoga or meditation within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Accrual Percentage--Persons with Dementia | Baseline
  Number of people randomized/Number of people approached about the study
Accrual Percentage--Caregivers | Baseline
  Number of people randomized/Number of people approached about the study
Percentage Adherence to Intervention Sessions--Persons with Dementia | Week 10
  Number of sessions attended/Total number of sessions offered
Percentage Adherence to Intervention Sessions--Caregivers | Week 10
  Number of sessions attended/Total number of sessions offered
Retention Percentage--Persons With Dementia | Week 10
  Number of people who complete the Week 10 assessment/Total Number Enrolled
Retention Percentage--Caregivers | Week 10
  Number of people who complete the Week 10 assessment/Total Number Enrolled

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire--Persons With Dementia | Week 10
  8-item measure of satisfaction with the intervention. Scores can range from 8 to 32; higher scores indicate more satisfaction.
Client Satisfaction Questionnaire--Caregivers | Week 10
  8-item measure of satisfaction with the intervention. Scores can range from 8 to 32; higher scores indicate more satisfaction.
Zarit Burden Interview | Baseline, Week 10
  Completed by caregiver. 22-item measure of caregiver burden. Scores range from 0 to 88, with higher scores indicating greater caregiver burden.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety--Persons with Dementia | Baseline, Week 10
  8-item measure of anxiety symptoms 8-item measure of anxiety symptoms; responses are made on a 5-point Likert scale and converted to t-scores with a mean of 50 and standard deviation of 10; higher scores indicate greater severity of anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety--Caregivers | Baseline, Week 10
  8-item measure of anxiety symptoms 8-item measure of anxiety symptoms; responses are made on a 5-point Likert scale and converted to t-scores with a mean of 50 and SD of 10; higher scores indicate greater severity of anxiety.
PROMIS Depression--Persons with Dementia | Baseline, Week 10
  8-item measure of depressive symptoms; responses are made on a 5-point Likert scale and converted to t-scores with a mean of 50 and SD of 10. higher scores indicate greater severity of depression.
PROMIS Depression--Caregivers | Baseline, Week 10
  8-item measure of depressive symptoms; responses are made on a 5-point Likert scale and converted to t-scores with a mean of 50 and SD of 10. higher scores indicate greater severity of depression.
PROMIS Self-efficacy for Managing Emotions--Persons with Dementia | Baseline, Week 10
  8-item measure of emotional regulation. Responses are made on a 5-point Likert scale and converted to t-scores with a mean of 50 and SD of 10 higher scores indicate greater self-efficacy.
PROMIS Self-efficacy for Managing Emotions--Caregivers | Baseline, Week 10
  8-item measure of emotional regulation. Responses are made on a 5-point Likert scale and converted to t-scores with a mean of 50 and SD of 10 higher scores indicate greater self-efficacy.
Neuropsychiatric Inventory Questionnaire--Severity | Baseline, Week 10
  Completed by caregivers. Severity and distress from 12 care recipient behavioral symptoms. Severity and distress from 12 care recipient behavioral symptoms are rated. Severity is rated on 3 point Likert scale and scores range from 12-36, with higher scores indicating greater severity.
Neuropsychiatric Inventory Questionnaire--Distress | Baseline, Week 10
  Completed by caregivers. Severity and distress from 12 care recipient behavioral symptoms. Severity and distress from 12 care recipient behavioral symptoms are rated. Distress is rated on a 6 point Likert scale and scores range from 0 to 60, with higher scores indicating greater distress
Insomnia Sleep Index--Persons with Dementia | Baseline, Week 10
  7-item self-report measure of type and severity of insomnia symptoms. 7-item measure of type and severity of insomnia symptoms; responses are made on a 5-point Likert scale and summed, with higher scores indicating greater insomnia; scores range from 0 to 28
Insomnia Sleep Index--Caregivers | Baseline, Week 10
  7-item self-report measure of type and severity of insomnia symptoms. 7-item measure of type and severity of insomnia symptoms; responses are made on a 5-point Likert scale and summed, with higher scores indicating greater insomnia; scores range from 0 to 28

OTHER OUTCOMES:
Percentage Adherence to Independent Practice--Persons With Dementia | Week 10
  Number of sessions of independent practice/Total number of recommended independent practice sessions (4X/week)
Percentage Adherence to Independent Practice--Caregivers | Week 10
  Number of sessions of independent practice/Total number of recommended independent practice sessions (4X/week)
Qualitative Questions | Baseline, Week 10
  Completed by caregivers. Any changes they noticed, motivation for engaging in yoga, barriers. Interview responses will be reviewed and common themes will be extracted.
Average Minutes of Yoga Practice per Day--Persons With Dementia | From Baseline through Week 10
  Collected from self-reported yoga/stretching log
Average Minutes of Yoga Practice per Day--Caregivers | From Baseline through Week 10
  Collected from self-reported yoga/stretching log

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Brenes, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05103839/ICF_000.pdf